CLINICAL TRIAL: NCT01254695
Title: Improving the Efficacy of Sacral Nerve Stimulation for Fecal Incontinence by Alteration of Stimulation Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 004
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Fecal Incontinence
Keywords: Idiopathic Fecal Incontinence; Fecal Incontinence; Sacral Nerve Stimulation; Sacral Nerve Neuromodulation
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Standard settings (Active Comparator): Amplitude: Sensory threshold Frequency:14 Hz Pulse width 210 μsec
  Interventions: Device: Medtronic InterStim / InterStim II
- Experimental Setting 1 (Experimental): Amplitude: Sensory threshold Frequency:6.9 Hz Pulse width 210 μsec
  Interventions: Device: Medtronic InterStim / InterStim II
- Experimental setting 2 (Experimental): Amplitude: Sensory threshold Frequency:31 Hz Pulse width 210 μsec
  Interventions: Device: Medtronic InterStim / InterStim II
- Experimental setting 3 (Experimental): Amplitude: Sensory threshold Frequency:14 Hz Pulse width 330 μsec
  Interventions: Device: Medtronic InterStim / InterStim II
- Experimental setting 4 (Experimental): Amplitude: Sensory threshold Frequency:14 Hz Pulse width 90 μsec
  Interventions: Device: Medtronic InterStim / InterStim II

INTERVENTIONS:
Device: Medtronic InterStim / InterStim II — Standard stimulation (Amplitude: sensory threshold, frequency 14 Hz, Pulsewidth 210 microsec.) will be compared wiht experimental setting 1,2,3,4
  Other Names: Medtronic InterStim; Medtronic InterStim II

SUMMARY:
Faecal incontinence is a devastating condition affecting 2,2 to 5 % of the adult population. The magnitude of the problem is probably underestimated. Sacral nerve stimulation (SNS), has over the last decade given hope to patient failing conservative treatment. Some patient do not have optimal continence after SNS-therapy. This study aims to identify optimal stimulation parameters - that will improve the functional outcome of SNS-therapy thru a double blinded randomized cross-over study.

DETAILED DESCRIPTION:
Faecal incontinence is a devastating condition affecting daily living and has major influences on quality of life. Faecal incontinence affects 2,2 to 5 % of the adult population. The magnitude of the problem is probably underestimated, because most patients don't discuss this affliction with their general practitioner. A new treatment, SNS has over the last decade given new hope to these patients. But a group of these patients has minor effect of the treatment - despite a satisfactory test-stimulation period. This study aims to identify optimal stimulation parameters that will improve patient continence and quality of life. Four different stimulation parameters will be tested through a double blind, randomized crossover study - standard stimulation parameters (frequency: 14 Hz, pulse width 210 microsec.) will serve as control stimulation.

The study includes five arms that will be tested in a randomized order. Each arm will be tested for four weeks in which the patient fill in bowel habit diaries and standardized questionnaires. The first week in each period will not be evaluated - is serves as a wash-out period.

Before any pacemaker changes anorectal manometry and rectal filling tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Diagnosed with idiopathic faecal incontinence,incontinence with minor (≤60 degrees) sphincteric defects or incontinence following sphincter repair.
* Medtronic Interstim IPG(pacemaker)implanted for more than 6 months
* minimum one incontinence episodes pr. week during ongoing SNS-therapy

Exclusion Criteria:

* Colorectal surgery after IPG-implantation
* Pregnancy or breastfeeding
* Anal/perianal pain or discomfort
* Patients who are not deemed able to follow the planned testing program, including mental illness or mentally unstable patients
* Medication with known effects on gastrointestinal motility, thyroid disease, diabetes, coeliac, neurological disorders.
* Spinal cord injury
* Irritable Bowel Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Quality of life changes | Will be assessed every four weeks during a twenty-week period
  Quality of life will be recorded by means of Rockwood faecal incontinence quality of life score. A total of five evaluations will be made every fourth week in the twenty week protocol perioed.

SECONDARY OUTCOMES:
Number of incontinence episodes | Will be assessed every four weeks durring a twenty-week period
  Assess number of incontinence episodes, by means of bowel habit diary. Four week bowel habit diary will be evaluated five times during the twenty-week protocol perioed.
Days with faecal soiling | Will be assessed every four weeks during a twenty-week period
  By means of a four week bowel habit diary
Days with faecal urgency. | Will be assessed every four weeks during a twelve-week period
  By means of a four week bowel habit diary
Wexner incontinence score | Will be assessed every four weeks during a twenty-week period
St. Marks Incontinence score | Will be assessed every four weeks during a twenty-week period
Assess changes in anorectal volume and pressure with different pacemaker settings | Will be assessed every four weeks during a twenty-week period
  Resting, maximal anal sphincter pressure and rectal filling(first sensation, urge to defacate and maximal tolerabel volume(Air))pressure will be measured with different pacemaker settings. In total five evaluations will be made in the twenty week protocol perioed.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob k Jakobsen, MD., Principal Investigator — Anal Physiology Laboratory, Surgical Research Section 900, Aarhus University Hospital, Denmark
Locations (2):
- Anal Physiology Laboratory, Surgical Research Section 900, Aarhus University Hospital, Aarhus, Aarhus C, Denmark
- St. Marks Hospital, London, Harrow - Middlesex, United Kingdom

REFERENCES:
- [Derived] Duelund-Jakobsen J, Dudding T, Bradshaw E, Buntzen S, Lundby L, Laurberg S, Vaizey C. Randomized double-blind crossover study of alternative stimulator settings in sacral nerve stimulation for faecal incontinence. Br J Surg. 2012 Oct;99(10):1445-52. doi: 10.1002/bjs.8867. PMID 22961528